CLINICAL TRIAL: NCT04838275
Title: A Mobile Health Exercise Prescription to Enhance Effectiveness of Antifibrotic Therapy in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: IPF mHealth Exercise Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Mary Beth Brown, Associate Professor, University of Washington
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00012537
Record Dates: First submitted 2021-04-05; First posted 2021-04-09 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise Arm (Experimental): antifibrotic therapy + mHealth monitoring + 12-wk mHealth home exercise prescription
  Interventions: Behavioral: 12-week mHealth home exercise prescription
- Non-Exercise Arm (No Intervention): antifibrotic therapy + mHealth monitoring

INTERVENTIONS:
Behavioral: 12-week mHealth home exercise prescription — 3x/week home walking protocol, 2x/week resistance exercise program
  Arms: Exercise Arm

SUMMARY:
Patients with idiopathic pulmonary fibrosis (IPF) who are stable on antifibrotic therapy at least 3 months will be randomized to complete a 12-week home exercise intervention using an mHealth platform, plus a pre- and post-intervention monitoring period (4 weeks each) and in-person study assessments.

DETAILED DESCRIPTION:
Contemporary walk test endpoints in IPF trials may under-represent patient functional gains with antifibrotic therapy, which may be more effectively captured with long-term activity monitoring. Traditional pulmonary rehabilitation centers create a barrier to patient exercise accessibility and compliance, which is eliminated in a mobile health (mHealth) exercise training approach. In this study, 30 patients with IPF will be randomized into one of two arms. The exercise arm will receive a 12-week home exercise intervention using an mHealth platform plus pre- and post-intervention monitoring (4 weeks each). The non-exercise arm will be monitored for the same study duration. The primary end point is change from baseline in daily physical activity as a number of weekly exercise minutes qualifying as moderate to vigorous physical activity (MVPA), METS*minutes of exercise per week, and sedentary time minutes. Assessments will be performed primarily via in-person study visits at week 4 and week 16, as well as via daily recordings from mHealth monitoring devices.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-80 yrs at randomization
* Diagnosis of idiopathic pulmonary fibrosis (IPF), consistent with the ATS 2018 Guidelines
* Percent Forced Vital Capacity (%FVC) ≥50%
* Percent Carbon Monoxide Diffusing Capacity (%DLCO) ≥30%
* Willing and able to participate in an exercise regimen
* Ambulatory without the use of an assistive device
* Stable on antifibrotic therapy (pirfenidone or nintedanib) at least 3 months
* No changes in other medication for at least 4 wks before enrollment
* Must be able to read, write, and verbally communicate in English

Exclusion Criteria:

* Forced expiratory volume in one second (FEV1)/FVC ratio <0.7 after administration of bronchodilator at screening
* Expected to receive a lung transplant within 1 year from randomization or, for patients at sites in the United States, on a lung transplant waiting list at randomization
* Known explanation for interstitial lung disease
* History of asthma or chronic obstructive pulmonary disease
* Active infection
* Ongoing IPF treatments including investigational therapy, immunosuppresents (other than prednisone 20 mg daily and below) and cytokine modulating agents
* Participation in a supervised exercise program including pulmonary rehab within the previous 12 months
* History of unstable or deteriorating cardiac or pulmonary disease (other than IPF) within the previous 6 months
* Major orthopedic, psychiatric, neurological, or other conditions that would impair performance of the study exercise outcomes
* Require >5LPM supplemental O2 at rest
* Currently pregnant

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Daily Physical Activity | 20 weeks
  Daily activity as step counts, intensity (metabolic equivalents), and duration (METS*min) of activity to identify number of minutes spent in moderate-to-vigorous physical activity (MVPA) vs. sedentary time
Rates of recruitment, adherence, completion and adverse events | 20 weeks
  As indicators of intervention feasibility.

SECONDARY OUTCOMES:
Oxygen Saturation (SpO2) | 12 weeks
  To monitor pulse oximetry second-by-second during exercise
Cardiopulmonary Exercise Testing (CPET) | Week 4, Week 16
  To assess for peak oxygen consumption, peak watts, and time to peak, resting/ peak/recovery heart rate, resting and exercise SpO2, and other variables
Pulmonary Function Tests (PFT) with DLCO | Week 4, Week 16
  To assess lung volumes and capacities indicative of pulmonary function
Six Minute Walk Test (6MWT) | Week 4, Week 16
  To assess walking distance and oxygen desaturation during submaximal exercise
Seated Knee Extension Maximal Force and Fatigue Curve Test | Week 4, Week 16
  With computerized dynamometer (Noraxon)
Lower Extremity Power Test | Week 4, Week 16
  With computerized dynamometer and interfacing force platform (Noraxon)
Wall Squat Functional Strength Test | Week 4, Week 16
  Functional strength testing of the lower extremities
Borg Rating of Perceived Dyspnea Scale | 20 weeks
  Survey dyspnea at rest and during exertion on a likert scale, with a range of 0-10. Higher scores indicate more severe shortness of breath.
IPF-specific version of the St. George Respiratory Questionnaire (SGRQ-I) | Week 4, Week 16, Week 20
  An idiopathic pulmonary fibrosis-specific health-related quality of life (HRQL) questionnaire. Domain and total scores are transformed to a range of 0-100, with higher scores indicating more impaired HRQL.
King's Brief Interstitial Lung Disease (KBILD) Questionnaire | Week 4, Week 16, Week 20
  An interstitial lung disease-specific, health-related quality of life (HRQL) questionnaire. KBILD domain and total scores are transformed to a range of 0-100. Higher scores indicate less impaired HRQL. A score of 100 = best health state.
Plasma brain natriuretic peptide (BNP) | Week 4, Week 16
  An indicator of cardiac wall stress

CONTACTS AND LOCATIONS:
Overall Officials: Mary Beth Brown, PT, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No